CLINICAL TRIAL: NCT01540721
Title: A Single Dose PK Study Investigating the Extent of Paracetamol Absorption From Two Different Sustained Released Paracetamol Formulations
Brief Title: Pharmacokinetic Study Investigating the Extent of Paracetamol Absorption From a New Formulation of Paracetamol Compared With Panadol® Extend
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A2750605
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Subjects
Keywords: paracetamol; pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental paracetamol formulation (Experimental): Experimental formulation
  Interventions: Drug: Experimental paracetamol formulation
- Marketed paracetamol (Active Comparator): Marketed formulation
  Interventions: Drug: Marketed paracetamol

INTERVENTIONS:
Drug: Marketed paracetamol — marketed formulation
  Arms: Marketed paracetamol
Drug: Experimental paracetamol formulation — Experimental formulation
  Arms: Experimental paracetamol formulation

SUMMARY:
This study will evaluate the pharmacokinetic profiles of experimental formulations of paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* Good health with (in the opinion of the investigator) no clinically significant and relevant abnormalities of medical history or physical examination

Exclusion Criteria:

* Current (within 14 days of screening) or regular use of any prescription, over the counter (OTC) drugs including paracetamol/acetaminophen, herbal medicine or drug known to induce or inhibit hepatic drug metabolism, excluding prescription birth control, if applicable.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Bioavailability as measured by Area Under the Curve (AUC) in both fasted and fed state | baseline to 12 hours
Effect of food on the extent and rate of paracetamol absorption as measured by AUC and Cmax | baseline to 12 hours

SECONDARY OUTCOMES:
To assess descriptive pharmaokinetic characteristics (Tmax, T1/2, Cmax, AUC) | baseline to 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- MDS Pharma Services NEBRASKA, Lincoln, Nebraska, United States